CLINICAL TRIAL: NCT01916876
Title: A Randomised Controlled Trial of an Integrated Post-discharge Transitional Care Package for General Medical In-patients in Cape Town, South Africa
Brief Title: Impact of Medical Follow-up Discharge Package
Acronym: RECALL-CT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding shortage
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Jonathan Peter, Honorary Consultant, Department of Medicine, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UCT 148.2/2013
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Follow-up Study; Medical In-patients
Keywords: medical in-patients; follow-up care; developing country

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): At discharge, patients will be given a discharge plan by their attending caregiver as deemed appropriate.
- Integrative medical follow-up package (Other): At discharge, patients will receive a discharge plan by their attending caregiver.
  Thereafter, if randomised to this study arm they will receive the intervention as outlined elsewhere.
  "Integrated Medical Follow-up package"
  Interventions: Other: Integrated medical follow-up package

INTERVENTIONS:
Other: Integrated medical follow-up package — At discharge, patients will receive a discharge plan by their attending caregiver.
  1. On day 3 they will be contacted telephonically to:
     i) Discuss their discharge diagnosis and medications ii) Arrange specialist clinic follow-up booking for 2 weeks iii) Reemphasise drug compliance
  2. Reminders via SMS to attend there OPD appointment(s)
  3. Medical out-patient review at 2-weeks and 6 weeks if required
  4. Medical telephonic "hot-line" for advice
  Arms: Integrative medical follow-up package

SUMMARY:
The post discharge time is a vulnerable time for general medical in-patients, with high rates of adverse events that may cause unnecessary readmissions and even death. A recent study of 415 patients discharged from the general medical wards at Groote Schuur Hospital, demonstrated a very high 12 month mortality of 35%. The majority of these deaths were classified as "unexpected". The reasons for this were not further examined, but it was speculated, given the authors' knowledge of the public sector in Cape Town, that three related factors contribute significantly to this early mortality: i) a lack of continuity of care, with patients not necessarily accessing the primary care support treatment that they need or being able to access early post discharge follow-up (for example for anti-retroviral or anti-tuberculous care); ii) the inability of primary care to deal with the complex nature of the discharged patients, most whom have significant co-morbid disease; iii) A lack of optimisation of therapy for chronic disease after acute discharge.

The investigators hypothesise that an integrated post-discharge transitional care package, which includes an early medical specialist follow-up in the first 3 months after hospital discharge will decrease the 6- and 12-month mortality and re-admission rate amongst general medical hospital admissions in Cape Town, South Africa. Our study will compare an integrated package, suitable to implementation if effective, with current standard discharge packages.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for admission to general medical wards (including within hospital transfer e.g. ICU discharge)
2. >18 years and willing to give informed consent

Exclusion Criteria:

1. Patient admitted directly to intensive care unit
2. Patient refusing consent or <18 years old
3. Patients electively admitted
4. Patients without phone numbers who cannot provide any telephone contact details for a co-habitant, relative or neighbour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 12 months
  All cause 12-month mortality will be evaluated at 12-months post enrolment. Data on mortality will be acquired through telephonic patient/family contact and review of provincial death registry

SECONDARY OUTCOMES:
All cause mortality | 6 months
  6-month mortality will be evaluated in a similar way to 12-month mortality.
Hospital readmission rate | 12 months
  Readmission to secondary, tertiary hospitals or emergency units will be included.
Bartel index | 12 months
  The change in functional outcome between discharge and 12-months will be measured using the Bartel index.
Karnofsky performance score | 12 months
  Changes in functional outcomes will be assessed by measuring the change in Karnofsky performance scores between 12-months and pre-admission.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Peter, Principal Investigator — University of Cape Town
Locations (2):
- South Africa (2):
  - Groote Schuur Hospital, Cape Town
  - Victoria Hospital, Cape Town

REFERENCES:
- [Background] Stuart-Clark H, Vorajee N, Zuma S, Van Niekerk L, Burch V, Raubenheimer P, Peter JG. Twelve-month outcomes of patients admitted to the acute general medical service at Groote Schuur Hospital. S Afr Med J. 2012 May 23;102(6):549-53. doi: 10.7196/samj.5615. PMID 22668961